CLINICAL TRIAL: NCT01340976
Title: A Phase 1 Safety Study of LY2787106 in Patients With Cancer and Anemia
Brief Title: A Phase 1 Study of LY2787106 in Cancer and Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13131; I3S-MC-JABA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-28; First posted 2011-04-25 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Anemia
Keywords: Cancer Related Anemia
MeSH Terms: conditions — Anemia | interventions — LY2787106

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2787106 Dose Escalation (Experimental): Part A: Dose escalation starting at 0.3 milligram/kilogram (mg/kg), intravenously (IV), day one of up to three 21-day cycles.
  Interventions: Drug: LY2787106
- 10 mg/kg LY2787106 (Experimental): Part B: 10 mg/kg of LY2787106, administered IV, on day one of up to eight 7-day cycles. Participants who do not experience a stopping rule and who are felt to be benefiting during the defined treatment period may receive additional doses at the discretion of the investigator.
  Interventions: Drug: LY2787106
- 10 mg/kg LY2787106+Iron (Experimental): Part B: 10 mg/kg of LY2787106, administered IV, on day one of up to eight 7-day cycles with daily oral iron supplementation. Participants who do not experience a stopping rule and who are felt to be benefiting during the defined treatment period may receive additional doses at the discretion of the investigator.
  Interventions: Drug: LY2787106; Dietary Supplement: Iron Supplementation

INTERVENTIONS:
Drug: LY2787106 — Administered IV.
Dietary Supplement: Iron Supplementation — Administered orally.
  Arms: 10 mg/kg LY2787106+Iron

SUMMARY:
This study will evaluate the safety LY2787106 in participants with cancer and anemia. It will also evaluate when LY2787106 can improve anemia. This study has two parts: Part A is a dose escalation evaluation. Part B is an evaluation of LY2787106 at a defined dose given with and without iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of non-myeloid cancer (solid tumors, lymphomas or multiple myeloma) that is metastatic and/or incurable
* Have been treated with at least one systemic (oral, intravenous, or subcutaneous) anti-cancer therapy or regimen
* Have a hemoglobin of less than or equal to 11 grams/deciliter (g/dL)
* Have a hepcidin level of greater than or equal to 5 nanograms/milliliter (ng/mL)
* Have given written informed consent prior to any study-specific procedures
* Have adequate hematologic, hepatic, and renal organ function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Available for the duration of the study and willing to follow study procedures
* If male or female with reproductive potential: Must agree to use medically approved contraception during the trial and for 4 months following the last dose of study drug
* If female with child bearing potential: Have a negative serum pregnancy test
* Have an estimated life expectancy of greater than or equal to 12 weeks

Exclusion Criteria:

* Have received treatment in the previous 21 days with, or have not recovered fully from, a drug that has not received regulatory approval for any indication
* Have received erythropoiesis-stimulating agents in the previous 21 days or red blood cell transfusions in the previous 14 days, or in the investigator's opinion, likely to need red blood cell transfusion more frequently than every 21 days
* Have received parenteral iron supplementation within the prior 14 days
* Have a documented history of pure red cell aplasia, thalassemia major or sickle cell disease
* Have a history of cirrhosis or major organ transplantation
* QTc greater than 470 millisecond (msec)
* Have evidence of clinically significant hemolysis or bleeding
* Have a clinically significant systemic infection within 14 days of enrollment
* Have a suspected or confirmed history of hemochromatosis.
* Have other serious preexisting medical conditions (left to the discretion of the investigator)
* Have symptomatic central nervous system malignancy or metastasis (screening not required)
* Have acute or chronic leukemia
* Are a female who is pregnant or lactating
* Have a history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C (screening not required)
* Have received external beam radiotherapy to more than 25% of the bone marrow
* Have known clinically significant hypersensitivity to biologic agents
* Have received live vaccine(s) within 1 month of screening or with plans of doing that during the participation to the study
* Have a history of congestive heart failure with New York Heart Association (NYHA) Class greater than 2 (NYHA Class 1 and 2 are eligible), unstable angina or recent myocardial infarction (within 1 year prior to administration of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington

REFERENCES:
- [Derived] Vadhan-Raj S, Abonour R, Goldman JW, Smith DA, Slapak CA, Ilaria RL Jr, Tiu RV, Wang X, Callies S, Cox J, Tuttle JL, Lau YK, Roeland EJ. A first-in-human phase 1 study of a hepcidin monoclonal antibody, LY2787106, in cancer-associated anemia. J Hematol Oncol. 2017 Mar 21;10(1):73. doi: 10.1186/s13045-017-0427-x. PMID 28327200

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part B participants who received 8 weekly doses and discontinued treatment were considered completers.
Groups:
- Part A 0.3 Milligram Per Kilogram (mg/kg) LY2787106: Part A: Participants received 0.3 mg/kg, LY2787106 intravenously (IV), day 1 of up to three 21-day cycles.
- Part A 1.0 mg/kg LY2787106: Part A: Participants received 1.0 mg/kg, LY2787106, IV, day 1 of up to three 21-day cycles.
- Part A 3.0 mg/kg LY2787106: Part A: Participants received 3.0 mg/kg, LY2787106, IV, day 1 of up to three 21-day cycles.
- Part A 10.0 mg/kg LY2787106: Part A: Participants received 10.0 mg/kg, LY2787106, IV, day 1 of up to three 21-day cycles.
- Part B 10.0 mg/kg LY2787106: Part B: Participants received 10.0 mg/kg LY2787106, IV, on day 1 of up to eight 7-day cycles.
- Part B 10.0 mg/kg LY2787106+Iron: Part B: Participants received 10.0 mg/kg, LY2787106, IV, on day 1 of up to eight 7-day cycles with daily oral iron supplementation.
Period: Overall Study
Arm/Group | Part A 0.3 Milligram Per Kilogram (mg/kg) LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Started | 4 | 3 | 7 | 5 | 7 | 7
Received at Least 1 Dose of Study Drug | 4 | 3 | 7 | 5 | 7 | 7
Completed | 0 | 1 | 4 | 2 | 5 | 6
Not Completed | 4 | 2 | 3 | 3 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 1 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Dose Limiting Toxicity Stopping Rule | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other anemia treatment | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A 0.3 mg/kg LY2787106: Part A: Participants received 0.3 mg/kg, LY2787106, IV, day 1 of up to three 21-day cycles.
- Part B 10.0 mg/kg LY2787106: Part B: Participants received 10.0 mg/kg, LY2787106, IV, on day 1 of up to eight 7-day cycles.
- Total: Total of all reporting groups
Arm/Group | Part A 0.3 mg/kg LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron | Total
Number analyzed (Participants) | 4 | 3 | 7 | 5 | 7 | 7 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.3) | 76.7 (12.7) | 62.1 (13.4) | 63.2 (7.9) | 66.3 (9.2) | 62.7 (7.5) | 64.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 3 | 4 | 6 | 20
  Male | 2 | 2 | 3 | 2 | 3 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 7 | 5 | 6 | 7 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 2 | 2 | 7
  White | 4 | 3 | 5 | 3 | 5 | 5 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7 | 5 | 7 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Events
Description: Number of participants with one or more treatment emergent adverse event (TEAE) or any Serious AE (SAE). A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline to Study Completion (up to 5 Years)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Part B 10 mg/kg LY2787106: Part B: Participants received 10 mg/kg, LY2787106, IV, on day 1 of up to eight 7-day cycles.
- Part B 10 mg/kg LY2787106+Iron: Part B: Participants received 10 mg/kg, LY2787106, IV, on day 1 of up to eight 7-day cycles with daily oral iron supplementation.
Arm/Group | Part A 0.3 mg/kg LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10 mg/kg LY2787106 | Part B 10 mg/kg LY2787106+Iron
Number analyzed (Participants) | 4 | 3 | 7 | 5 | 7 | 7
participants
  Participants with at least 1 TEAE event | 4 | 3 | 6 | 5 | 0 | 0
  Participants with at least 1 SAE event | 1 | 2 | 2 | 0 | 0 | 1

2. Primary Outcome: Mean Change From Baseline in Hemoglobin With or Without Oral Iron Supplementation
Description: This analysis assesses the mean change in Hemoglobin from baseline to the end of Cycle 4. The analysis was carried separately for Cohort B1 without supplemental iron and Cohort B2 with supplemental iron.
Time Frame: Baseline, Cycle 4 (7-day cycle)
Population: Evaluable population in Part B is defined as a participant who received all 4 of the first 4 per-cycle doses of study medication, maintained at least 60% compliance with oral iron therapy during the first 4 cycles of LY2787106 (if enrolled to the oral iron cohort), and who had a hemoglobin assessment after each of the first 4 doses.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Part B 10 mg/kg LY2787106 | Part B 10 mg/kg LY2787106+Iron
Number analyzed (Participants) | 6 | 6
grams per deciliter (g/dL) | -0.5 (0.49) | -0.2 (0.80)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax)
Description: Cmax is the maximum serum concentration after a single IV dose of the study drug.
Time Frame: Days 1, 2, and 4 of Cycles 1 and 5, Day 1 of Cycles 2, 3, 4, 6, 7 and 8 (Part A 21-day cycles, Part B 7-day cycles) and 1, 3, and 9 weeks after the last infusion
Population: All participants who received at least 1 dose of study drug and who had evaluable PK data for Cmax.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Part A 0.3 mg/kg LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Number analyzed (Participants) | 4 | 3 | 7 | 5 | 5 | 6
nanogram per milliliter (ng/ml) | 5450 (24) | 22300 (27) | 79000 (15) | 205000 (12) | 258000 (15) | 199000 (12)

4. Secondary Outcome: PK: Area Under the Curve (AUC[0-∞])
Description: AUC is the area under the concentration versus time curve from time zero to infinity.
Time Frame: as for outcome 3
Population: All participants who received at least 1 dose of study drug and who had evaluable PK data for AUC[0-∞]).
Measure: Mean (Standard Deviation); unit: micrograms∙hour per milliliter (µg∙h/mL)
Arm/Group | Part A 0.3 mg/kg LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Number analyzed (Participants) | 4 | 3 | 7 | 5 | 6 | 5
micrograms∙hour per milliliter (µg∙h/mL) | 663 (42) | 2146 (64) | 8934 (39) | 24503 (19) | 21000 (19) | 16798 (27)

5. Secondary Outcome: Recommended Dose for Future Studies: Maximum Tolerated Dose (MTD)
Description: MTD is defined as being the highest tested dose below the level at which one-third or more of participants experience a Dose-limiting toxicity (DLT). DLT is defined as an adverse event occurring in any part of the study that is related to the study medication, occurs during Cycle 1 of Part A, and fulfills any one of the following criteria:
  1. Clinically significant Grade 2 toxicity, such as angina, arrhythmia, seizure, dyspnea, rash with significant blistering or desquamation, or other event deemed significant by either the investigator.
  2. ≥Grade 3 anemia (excluding participants with baseline <9.0 g/dL) or hemoglobin (Hb) decrease >1.0 g/dL if baseline Hb <9.0 g/dL, confirmed by 2 independent measurements.
  3. ≥ Grade 3 cytokine release syndrome/acute infusion reaction.
  4. Other ≥ Grade 3 hematological or non-hematological toxicity.
Time Frame: Baseline to Cycle 1 of Part A
Population: MTD was not determined in this study, so zero participants were analyzed.
Arm/Group | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Serum Iron
Description: Mean change in serum iron from baseline to the end of Cycle 4.
Time Frame: Baseline, Cycle 4 (7-day cycle)
Population: Evaluable Population in Part B is defined as a participant who has received all 4 of the first 4 per-cycle doses of study dose, maintained at least 60% compliance with oral iron therapy during the first 4 cycles of LY2787106 (if enrolled to the oral iron cohort), and who has had a hemoglobin assessment after each of the first 4 doses.
Measure: Mean (Standard Deviation); unit: micromole per liter (umol/L)
Arm/Group | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Number analyzed (Participants) | 6 | 6
micromole per liter (umol/L) | -0.4 (6.17) | -4.6 (9.20)

7. Secondary Outcome: Mean Change From Baseline in Reticulocyte Count
Description: Mean change in reticulocyte count from baseline to the end of Cycle 4.
Time Frame: Baseline, Cycle 4 (7-day cycle)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of reticulytes
Arm/Group | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Number analyzed (Participants) | 4 | 6
percentage of reticulytes | 1.2 (0.68) | 0.0 (0.46)

ADVERSE EVENTS:
Groups:
- Part B 10.0 mg/kg LY2787106: Part B: Participants received 10.0 mg/kg of LY2787106, administered IV, on day 1 of up to eight 7-day cycles.
- Part B 10.0 mg/kg LY2787106+Iron: Part B: 10.0 mg/kg, LY2787106, IV, on day 1 of up to eight 7-day cycles with daily oral iron supplementation.
Arm/Group | Part A 0.3 mg/kg LY2787106 | Part A 1.0 mg/kg LY2787106 | Part A 3.0 mg/kg LY2787106 | Part A 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106 | Part B 10.0 mg/kg LY2787106+Iron
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/3 | 2/7 | 0/5 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/7 | 5/5 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A 0.3 mg/kg LY2787106 (N=4) | Part A 1.0 mg/kg LY2787106 (N=3) | Part A 3.0 mg/kg LY2787106 (N=7) | Part A 10.0 mg/kg LY2787106 (N=5) | Part B 10.0 mg/kg LY2787106 (N=7) | Part B 10.0 mg/kg LY2787106+Iron (N=7)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A 0.3 mg/kg LY2787106 (N=4) | Part A 1.0 mg/kg LY2787106 (N=3) | Part A 3.0 mg/kg LY2787106 (N=7) | Part A 10.0 mg/kg LY2787106 (N=5) | Part B 10.0 mg/kg LY2787106 (N=7) | Part B 10.0 mg/kg LY2787106+Iron (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 3 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (10) | 4 (6)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (4) | 2 (4) | 0 (0) | 5 (25) | 7 (35)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Genital abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (34) | 1 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (8)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (18) | 2 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (18) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0/2 (0) | 0/1 (0) | 0/4 (0) | 1/3 (1) | 0/4 (0) | 0/6 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days